CLINICAL TRIAL: NCT06154434
Title: An Open Label, Randomized, Fasting, Single-dose, Two-period Crossover Study to Compare the Bioequivalence of Chlorpromazine HCl 100mg Tablets After Oral Administration in Healthy Subjects.
Brief Title: Bioequivalence Study in Healthy Subjects by Using of Chlorpromazine HCl 100mg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Whanin Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DDS16-065BE
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Healthy Subject
MeSH Terms: interventions — Chlorpromazine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: Chlorpromazine HCl 100mg Tablets
- Group B (Experimental)
  Interventions: Drug: Chlorpromazine HCl 100mg Tablets

INTERVENTIONS:
Drug: Chlorpromazine HCl 100mg Tablets — single-dose administered after a 10-hour overnight fast.

SUMMARY:
This clinical study is an open label, randomized, fasting condition, single-dose, two-period crossover study to compare the bioequivalence of Chlorpromazine HCl 100mg Tablets after oral administration in healthy subjects.

ELIGIBILITY:
Main Inclusion Criteria:

1. Healthy subjects, over the age of 19 years old
2. Weight: At least 50.0 kg and Body mass index (BMI) between 18.0-30.0 kg/m2.
3. All subjects should be judged normal and healthy during a pre-study medical evaluation

   * Subjects who has no birth or chronic disease and must be in good health as determined by physical exmination and medical tests including biochemistry, urinalysis, serology and hematology etc in serum/urine.
4. Subject is willing to participate and to Sign written informed consent form
5. Female subjects of childbearing age who use contraception other than hormonal contraception.
6. Subjects who has no history of psychical disorder within the last five years

Main Exclusion Criteria:

1. Subjects who have a medical history specified in protocol
2. Subjects who are expected to have the prohibited medication and activity etc. during the study period
3. Subjects who can not comply with requirements as per protocol
4. Pregnant women or breast-feeding women or men and women who has possibility of pregnancy
5. Subjects who are not suitable for the clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
AUClast | Up to 72 hours
Cmax | Up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: MINGYU PARK, Principal Investigator — Chungbuk National University Hospital
Locations (1):
- Whan In Pharm., Seoul, South Korea